CLINICAL TRIAL: NCT02018536
Title: A Phase 1, Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of GSK2336805 (Part 1), Followed by an Open-label, Randomized, 4-way Crossover Study to Evaluate Short-term Safety, Tolerability and Pharmacokinetics of the Co-administration of TMC435 and GSK2336805 at Steady-state (Part 2), in Healthy Japanese Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK2336805 Alone and With the Co-administration of TMC435 in Healthy Japanese Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR102928; TMC435HPC1012 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Healthy; TMC435; GSK2336805; Pharmacokinetic; Safety; Tolerability
MeSH Terms: interventions — GSK2336805; Simeprevir; Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1, Cohort A (Experimental): 8 participants to receive a single oral dose of 30 mg of GSK2336805 (6 participants) or placebo (2 participants) on Day 1.
  Interventions: Drug: GSK2336805 30 mg
- Part 1, Cohort B (Experimental): 8 participants to receive a single oral dose of 60 mg of GSK2336805 (6 participants) or placebo (2 participants) on Day 1.
  Interventions: Drug: GSK2336805 60 mg
- Part 1, Cohort C (Experimental): 8 participants to receive a single oral dose of 120 mg of GSK2336805 (6 participants) or placebo (2 participants) on Day 1.
  Interventions: Drug: GSK2336805 120 mg
- Part 2, Sequence 1 (Experimental): 6 participants to receive Treatment A (TMC435 150 mg), D (TMC435 150 mg+GSK2336805 60 mg), B (GSK2336805 60 mg), and C (TMC435 100 mg+GSK2336805 60 mg) in a sequence with a 7 days washout period between each treatment sessions.
  Interventions: Drug: TMC435 150 mg (Treatment A); Drug: GSK2336805 60 mg (Treatment B and part of Treatment C and D); Drug: TMC435 100 mg (part of Treatment C); Drug: TMC435 150 mg (part of treatment D)
- Part 2, Sequence 2 (Experimental): 6 participants to receive Treatment B (GSK2336805 60 mg), A (TMC435 150 mg), C (TMC435 100 mg+GSK2336805 60 mg), and D (TMC435 150 mg+GSK2336805 60 mg) in a sequence with a 7 days washout period between each treatment sessions.
  Interventions: Drug: TMC435 150 mg (Treatment A); Drug: GSK2336805 60 mg (Treatment B and part of Treatment C and D); Drug: TMC435 100 mg (part of Treatment C); Drug: TMC435 150 mg (part of treatment D)
- Part 2, Sequence 3 (Experimental): 6 participants to receive Treatment C (TMC435 100 mg+GSK2336805 60 mg), B (GSK2336805 60 mg), D (TMC435 150 mg+GSK2336805 60 mg), and A (TMC435 150 mg) in a sequence with a 7 days washout period between each treatment sessions.
  Interventions: Drug: TMC435 150 mg (Treatment A); Drug: GSK2336805 60 mg (Treatment B and part of Treatment C and D); Drug: TMC435 100 mg (part of Treatment C); Drug: TMC435 150 mg (part of treatment D)
- Part 2, Sequence 4 (Experimental): 6 participants to receive Treatment D (TMC435 150 mg+GSK2336805 60 mg), C (TMC435 100 mg+GSK2336805 60 mg), A (TMC435 150 mg) and B (GSK2336805 60 mg) in a sequence with a 7 days washout period between each treatment sessions.
  Interventions: Drug: TMC435 150 mg (Treatment A); Drug: GSK2336805 60 mg (Treatment B and part of Treatment C and D); Drug: TMC435 100 mg (part of Treatment C); Drug: TMC435 150 mg (part of treatment D)

INTERVENTIONS:
Drug: GSK2336805 30 mg — A single dose of 1 tablet of 30 mg of GSK2336805 taken orally (by mouth) on Day 1 under fasted conditions.
  Arms: Part 1, Cohort A
Drug: GSK2336805 60 mg — A single dose of 2 tablets of 30 mg ie, 60 mg of GSK2336805 taken orally (by mouth) on Day 1 under fasted conditions.
  Arms: Part 1, Cohort B
Drug: GSK2336805 120 mg — A single dose of 4 tablets of 30 mg ie, 120 mg of GSK2336805 taken orally (by mouth) on Day 1 under fasted conditions.
  Arms: Part 1, Cohort C
Drug: TMC435 150 mg (Treatment A) — 1 capsule of TMC435 150 mg taken once daily orally (by mouth) on Days 1 to 7 under fed conditions.
  Arms: Part 2, Sequence 1; Part 2, Sequence 2; Part 2, Sequence 3; Part 2, Sequence 4
Drug: GSK2336805 60 mg (Treatment B and part of Treatment C and D) — 2 tablets of 30 mg GSK2336805 ie, 60 mg of GSK2336805 taken once daily orally (by mouth) on Days 1 to 7 under fed conditions.
  Arms: Part 2, Sequence 1; Part 2, Sequence 2; Part 2, Sequence 3; Part 2, Sequence 4
Drug: TMC435 100 mg (part of Treatment C) — 1 capsule of TMC435 100 mg taken orally (by mouth) on Days 1 to 7 under fed conditions.
  Arms: Part 2, Sequence 1; Part 2, Sequence 2; Part 2, Sequence 3; Part 2, Sequence 4
Drug: TMC435 150 mg (part of treatment D) — 1 capsule of TMC435 150 mg taken orally (by mouth) on Days 1 to 7 under fed conditions.
  Arms: Part 2, Sequence 1; Part 2, Sequence 2; Part 2, Sequence 3; Part 2, Sequence 4

SUMMARY:
The purpose of the study is to investigate the safety, tolerability, and pharmacokinetic (what the body does to a medication) of GSK2336805 alone and with the co-administration of TMC435 in healthy Japanese participants.

DETAILED DESCRIPTION:
This study will consists of 2 parts (Part 1 and 2) which will be sequentially conducted in 2 separate panels of 24 healthy adult Japanese participants each, at a single center. Part 1 is a double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (placebo is compared with the study medication to test whether the study medication has a real effect in clinical study), randomized (study medication is assigned by chance), single ascending dose study to investigate the safety, tolerability, and pharmacokinetics of GSK2336805 in participants. It will consist of a screening phase, a treatment phase, and a follow-up phase. The maximum study duration for each participant will be approximately 5 weeks (including screening and follow-up phase). 24 participants will be equally divided in 3 cohorts with 8 participants in each cohort. In each cohort, participants will be randomly assigned to receive either a single oral dose of GSK2336805 (6 participants) or placebo (2 participants). Part 2 is an open-label (all people know the identity of the intervention), randomized, 4-way crossover study (method used to switch patients from one treatment arm to another in a clinical study) to investigate the potential pharmacokinetic drug-drug interactions between TMC435 and GSK2336805 at steady-state, and to evaluate the short-term safety and tolerability when TMC435 and GSK2336805 are co-administered in participants. It will consist of a screening phase, a treatment phase (4 treatment sessions [Treatment A, B, C, and D]), and a follow-up phase. The maximum study duration for each participant will be approximately 12 weeks (including screening and follow-up phase). During 4 treatment sessions, each of the 24 participants will receive Treatment A, B, C and D consecutively in different sequences with a washout period of at least 7 days between consecutive treatment sessions in each individual participant. Safety will be evaluated by assessing adverse events, clinical laboratory tests, electrocardiogram, vital signs, physical examination, alcohol breath tests, and specific toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese participants on the basis of medical history, physical examination, vital signs, triplicate 12-lead electrocardiogram, and clinical laboratory testing performed at screening
* Must have signed an Informed Consent Form (ICF) indicating they understand the purpose of and procedures required for the study
* Must be willing to adhere to the prohibitions and restrictions specified in the protocol
* Women must be of non-childbearing potential (postmenopausal for at least 2 years or surgically sterile)
* Women, except for postmenopausal women, should have a negative serum b-human chorionic gonadotropin (hCG) pregnancy test at screening

Exclusion Criteria:

* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use within the past one year
* Participants with hepatitis A, B, or C infection or human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection at study screening
* Female participants who are breastfeeding at screening
* History of liver or renal impairment; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Participants with known allergies, hypersensitivity, or intolerance to GSK2336805, TMC435 or excipients of the drug products used

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum observed plasma concentration of GSK2336805 | Predose, postdose on Day 1 (0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours), Day 2 (24 and 36 hour), Day 3, and time point of early withdrawal
Part 1: Area under the plasma concentration-time curve of GSK2336805 | Predose, postdose on Day 1 (0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours), Day 2 (24 and 36 hour), Day 3, and time point of early withdrawal
Part 1: The actual sampling time to reach the maximum observed plasma concentration of GSK2336805 | Predose, postdose on Day 1 (0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours), Day 2 (24 and 36 hour), Day 3, and time point of early withdrawal
Part 2: Maximum observed plasma concentration of TMC435 | Predose, postdose on Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 2, Day 5, Day 6, Day 7 (predose and postdose (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 8, Day 9, Day 10, and time point of early withdrawal
Part 2: Area under the plasma concentration-time curve of TMC435 | Predose, postdose on Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 2, Day 5, Day 6, Day 7 (predose and postdose (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 8, Day 9, Day 10, and time point of early withdrawal
Part 2: The actual sampling time to reach the maximum observed plasma concentration of TMC435 | Predose, postdose on Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 2, Day 5, Day 6, Day 7 (predose and postdose (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 8, Day 9, Day 10, and time point of early withdrawal
Part 2: Maximum observed plasma concentration of GSK2336805 | Predose, postdose on Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 2, Day 5, Day 6, Day 7 (predose and postdose (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 8, Day 9, Day 10, and time point of early withdrawal
Part 2: Area under the plasma concentration-time curve of GSK2336805 | Predose, postdose on Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 2, Day 5, Day 6, Day 7 (predose and postdose (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 8, Day 9, Day 10, and time point of early withdrawal
Part 2: The actual sampling time to reach the maximum observed plasma concentration of GSK2336805 | Predose, postdose on Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 2, Day 5, Day 6, Day 7 (predose and postdose (0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours), Day 8, Day 9, Day 10, and time point of early withdrawal

SECONDARY OUTCOMES:
Part 1 and 2: Number of participants with adverse events | Up to 12-14 weeks
  Number of participants with adverse events as a measure of safety and tolerability after administration of TMC435 alone, GSK2336805 alone, and after TMC435 administration in combination with GSK2336805

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Cypress, California, United States